CLINICAL TRIAL: NCT06553183
Title: Immersive Virtual Reality Based Exersice and Shoulder Proprioception and Range of Motion in Post-mastectomy Lymphedema Patients
Brief Title: Immersive Virtual Reality Based Exersice in Post-mastectomy Lymphedema Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, doaa atef, lecturer of physical therapy for surgery, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/005255
Record Dates: First submitted 2024-08-08; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Lymphedema Arm

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): the patients will receive eight sessions of Immersive virtual reality based exercise, 2 sessions per week for 4 weeks besides the traditional physical therapy.
  Interventions: Procedure: immersive virtual reality; Procedure: traditional physicaltherapy
- control group (Active Comparator): the patients will receive eight sessions of the traditional physical therapy, 2 sessions per week for 4 weeks.
  Interventions: Procedure: traditional physicaltherapy

INTERVENTIONS:
Procedure: immersive virtual reality — Exercise based on virtual reality video games. Immersive type will be used.
  Arms: study group
Procedure: traditional physicaltherapy — pneumatic compression, exercise and skin care

SUMMARY:
To determine the effect of immersive virtual reality on shoulder proprioception and ROM of post-mastectomy lymphedema patients.

DETAILED DESCRIPTION:
RESEARCH QUESTION:

Does Immersive virtual reality based exercise effective in improving shoulder proprioception and ROM for post-mastectomy patients?

Assessment:

The digital goniometer will be used in measuring shoulder extension, flexion, adduction, abduction, internal rotation and external rotation before the sessions and after one month of sessions. Also, shoulder proprioception will be assessed by the digital goniometer.The measurement will be taken for both the edematous side and the non-affected side.

Treatment:

Study group: the patients will receive eight sessions of Immersive virtual reality based exercise, 2 sessions per week for 4 weeks besides the traditional physical therapy.

Control group: the patients will receive eight sessions of the traditional physical therapy, 2 sessions per week for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* All the patients will be females.
* Patients with lymph node dissection.
* start at least 2 weeks after operation.

Exclusion Criteria:

* Vision problems.
* Medically instable patients.
* Balance disorders.
* Other musculoskeletal condition of shoulders.

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-15 (Estimated); Primary Completion 2025-01-15 (Estimated); Study Completion 2025-02-15 (Estimated)

PRIMARY OUTCOMES:
shoulder proprioception | 4 weeks
  digital goniometer

SECONDARY OUTCOMES:
shoulder ROM | 4 weeks
  all 6 motions will be measured by digital goniometer

IPD SHARING:
Plan to Share IPD: No